CLINICAL TRIAL: NCT03039036
Title: A Randomized Clinical Trial of Early Amniotomy Versus Delayed Amniotomy Following Foley Catheter Ripening in Nulliparous Labor Induction
Brief Title: Early Amniotomy Versus Delayed Amniotomy Following Foley Catheter Ripening in Nulliparous Labor Induction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Emily Miller, Assistant Professor of Obstetrics and Gynecology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00204292
Record Dates: First submitted 2016-12-15; First posted 2017-02-01 (Estimated); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Labor Induction
Keywords: Labor Induction; Early Amniotomy; Foley catheter
MeSH Terms: interventions — Amniotomy; Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Amniotomy (Experimental): Patients undergoing induction of labor with foley catheter, with or without concurrent use of misoprostol, will undergo amniotomy within 1 hour of Foley catheter removal.
  Interventions: Procedure: Amniotomy; Device: Foley Catheter; Drug: Misoprostol
- Delayed Amniotomy (Active Comparator): Patients undergoing induction of labor with foley catheter, with or without concurrent use of misoprostol, will undergo amniotomy no sooner than 4 hours following removal of Foley catheter.
  Interventions: Procedure: Amniotomy; Device: Foley Catheter; Drug: Misoprostol

INTERVENTIONS:
Procedure: Amniotomy — Artificially rupturing membranes
Device: Foley Catheter — Foley catheter device is commonly used for cervical ripening during labor induction. It is used independently or in combination with pharmacologic augmentation. It is inserted in the cervix and the balloon is then inflated with 60 cc of saline. It is removed when either 1. it falls out under gentile traction during labor checks or 2. it is de-inflated at 12 hours after placement. If at the time of de-inflation at 12 hours, the desired affect has not been achieved, the provider may choose to place another foley balloon or use an alternative method of induction (misoprostol). This is an eligibility criteria and only patients who are undergoing induction with a Foley Catheter will be approached for enrollment.
Drug: Misoprostol — Misoprostol is a medication that is commonly used for cervical ripening during labor induction. It is commonly used independently or in combination with mechanical methods, such as a foley catheter. The commonly used dose during term labor induction is 25 mcg. Use of this medication will be decided by the provider.

SUMMARY:
Amniotomy (breaking the bag of water) is commonly used in the induction of labor. However, the timing is highly variable. The purpose of this study is to determine if first time mothers undergoing induction of labor with a Foley catheter experience a decrease in their labor time when undergoing early amniotomy (breaking the bag of water within 1 hour of Foley catheter removal) than when undergoing delayed amniotomy (breaking the bag of water at least 4 hours after Foley catheter removal). Other aims include the relationship between timing of amniotomy and cesarean section, postpartum hemorrhage, intrauterine infection, neonatal Apgar score <7 at 5 minutes, neonatal need for intensive care.

The investigators hypothesize that induction of labor with Foley catheters followed by early amniotomy will result in a decreased duration of labor compared to those who undergo delayed amniotomy.

DETAILED DESCRIPTION:
This randomized clinical trial of consenting nulliparous women undergoing induction of labor with a Foley catheter seeks to determine whether use of early amniotomy (defined as amniotomy within 1 hour of Foley catheter removal) improves obstetrical outcomes when compared with delayed amniotomy (defined as amniotomy at least 4 hours following Foley catheter removal).

This project will include 110 women recruited from the obstetrical service at Prentice Women's Hospital. Women will be included if they are at least 37 weeks gestation, have a singleton pregnancy, have intact membranes and are undergoing an induction of labor using a Foley catheter. Following removal of Foley catheter, women will be assessed for safety of amniotomy and if appropriate, randomized to either early amniotomy or delayed amniotomy.

Women will be randomized with equal probability to the intervention group using block randomization stratified by use of Foley catheter alone or Foley catheter-misoprostol use.

Women in the early amniotomy group will undergo amniotomy within 1 hour of Foley catheter removal. Women in the delayed amniotomy group will undergo amniotomy at least 4 hours following Foley removal. The remainder of labor management will be at the discretion of each woman's obstetric provider.

Prior to discharge from the hospital, baseline demographic and clinical data will be obtained via chart review

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* English speaking
* Women age 18 years old or greater
* Nulliparous
* Pregnant with a singleton gestation that is greater than or equal to 37 weeks
* Undergoing induction of labor with Foley catheter

Exclusion Criteria:

* Women not meeting above criteria
* Fetus in non-cephalic position
* Intrauterine fetal demise
* Fetus with major anomalies
* HIV, hepatitis B or C infection
* Planned use of oxytocin during the Foley catheter ripening

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Time interval from Foley catheter removal to delivery | Number of hours from removal of Foley catheter to delivery of neonate; up to 72 hours.
  Hours

SECONDARY OUTCOMES:
Cesarean delivery | At time of delivery
  binary; yes/no
Chorioamnionitis | From time of admission to Labor and Delivery unit to delivery of neonate; up to 72 hours
  Maternal Temperature of >/= 39 degrees Celsius or >/= 38 degrees Celsius on two occasions greater than 30 minutes apart and at least one of the following: Fetal tachycardia (defined as sustained (>10 min) fetal heart rate >160), White Bood Cell Count >15, purulent fluid from cervical os, or receipt of antibiotics and diagnosis written in the chart
Postpartum Fever | From time of delivery to time of hospital discharge; up to 6 weeks
  Temperature >/= 38 degrees celsius on 2 separate occasions greater than 6 hours apart
Wound infection | From time of delivery to time of hospital discharge; up to 6 weeks
  Cellulitis or erythema and induration around the incision and purulent discharge from the incision site with or without fever
Endometritis | From time of delivery to time of hospital discharge; up to 6 weeks
  fundal tenderness and fever that required treatment with antibiotics
5 minute Apgar Score less than 7 out of 10 | 5 minutes following delivery; 5 minutes of neonatal life.
  Neonatal Apgar scores consist of measurements of neonatal skin color, respiratory rate, heart rate, muscle tone, and irritability. Each parameter is given a score of 0, 1 or 2 based on standardized parameters. It is standard to perform this on all neonates at 1 minute and 5 minutes of life. Apgar scores are performed and calculated by nursing staff or members of the pediatric team. For this outcome, we are interested in scores less than 7 out of 10 at 5 minutes of life.
Neonatal intensive care unit admission | From time of delivery to hospital discharge; up to 6 weeks
  Admission to the neonatal intensive care unit for greater than 24 hours
Length of Labor | Time from placement of Foley catheter to time of delivery of neonate; up to 5 days
  hours
Suspected or confirmed neonatal sepsis | From time of delivery to hospital discharge; up to 6 weeks
  As clinical suspected by the neonatology team or with positive cultures
Postpartum hemorrhage | From time of delivery to time of hospital discharge; up to 6 weeks
  Delivery estimated blood loss of > 500 cc for vaginal delivery or > 1000 cc for cesarean delivery
Delivery time less than 24 hours | From time of placement of Foley catheter to time of delivery of neonate; within 24 hours.
  binary; yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Emily Miller, MD, Principal Investigator — Northwestern University
Locations (1):
- Prentice Women's Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Osterman MJ, Martin JA. Recent declines in induction of labor by gestational age. NCHS Data Brief. 2014 Jun;(155):1-8. PMID 24941926
- [Background] Maslow AS, Sweeny AL. Elective induction of labor as a risk factor for cesarean delivery among low-risk women at term. Obstet Gynecol. 2000 Jun;95(6 Pt 1):917-22. doi: 10.1016/s0029-7844(00)00794-8. PMID 10831992
- [Background] Garcia-Simon R, Montanes A, Clemente J, Del Pino MD, Romero MA, Fabre E, Oros D. Economic implications of labor induction. Int J Gynaecol Obstet. 2016 Apr;133(1):112-5. doi: 10.1016/j.ijgo.2015.08.022. Epub 2015 Dec 18. PMID 26868065
- [Background] Carbone JF, Tuuli MG, Fogertey PJ, Roehl KA, Macones GA. Combination of Foley bulb and vaginal misoprostol compared with vaginal misoprostol alone for cervical ripening and labor induction: a randomized controlled trial. Obstet Gynecol. 2013 Feb;121(2 Pt 1):247-252. doi: 10.1097/AOG.0b013e31827e5dca. PMID 23303106
- [Background] Smyth RM, Markham C, Dowswell T. Amniotomy for shortening spontaneous labour. Cochrane Database Syst Rev. 2013 Jun 18;2013(6):CD006167. doi: 10.1002/14651858.CD006167.pub4. PMID 23780653
- [Background] Gelber S, Sciscione A. Mechanical methods of cervical ripening and labor induction. Clin Obstet Gynecol. 2006 Sep;49(3):642-57. doi: 10.1097/00003081-200609000-00022. PMID 16885669
- [Background] Jozwiak M, Bloemenkamp KW, Kelly AJ, Mol BW, Irion O, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2012 Mar 14;(3):CD001233. doi: 10.1002/14651858.CD001233.pub2. PMID 22419277
- [Background] Mizrachi Y, Levy M, Bar J, Kovo M. Induction of labor in nulliparous women with unfavorable cervix: a comparison of Foley catheter and vaginal prostaglandin E2. Arch Gynecol Obstet. 2016 Oct;294(4):725-30. doi: 10.1007/s00404-016-4026-9. Epub 2016 Feb 2. PMID 26837386
- [Background] Levy R, Ferber A, Ben-Arie A, Paz B, Hazan Y, Blickstein I, Hagay ZJ. A randomised comparison of early versus late amniotomy following cervical ripening with a Foley catheter. BJOG. 2002 Feb;109(2):168-72. doi: 10.1111/j.1471-0528.2002.01137.x. PMID 11888099
- [Background] Battarbee AN, Palatnik A, Peress DA, Grobman WA. Association of Early Amniotomy After Foley Balloon Catheter Ripening and Duration of Nulliparous Labor Induction. Obstet Gynecol. 2016 Sep;128(3):592-597. doi: 10.1097/AOG.0000000000001563. PMID 27500341
- [Background] Levine LD, Downes KL, Elovitz MA, Parry S, Sammel MD, Srinivas SK. Mechanical and Pharmacologic Methods of Labor Induction: A Randomized Controlled Trial. Obstet Gynecol. 2016 Dec;128(6):1357-1364. doi: 10.1097/AOG.0000000000001778. PMID 27824758